CLINICAL TRIAL: NCT06129383
Title: The Effect of Adding Pectointercostal Plane Block to Serratus Anterior Plane Block on Postoparative Pain Management in Patient Planned for Breast Surgery
Brief Title: The Effect of Adding PIFP Block to SAP Block on Postoparative Pain Management in Patient Planned for Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Özlem Gök, DOCTOR, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-16/7
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pain Management
Keywords: Pecto-intercostal facial block; breast surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Within the scope of this study, two different research groups were identified for which clinical research was planned. The significance level of the power analysis was determined as 0.05 and the power level was determined as 0.80. However, for this study, it was decided to consider the effect size value as 0.4, based on similar studies in the literature. It was deemed sufficient to include n = 26 cases in each group, and it was deemed appropriate to include n = 30 cases in each group, considering a 20% wastage margin. The cases will be divided into 2 groups of 30 people using the sealed envelope method. Group I will include patients who underwent SAP block under general anesthesia (Control group), and Group II will include patients who underwent SAP and PIFB block under general anesthesia (Experimental group).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group to which serratus anterior plane block will be applied (Active Comparator): Control group patients, accompanied by the 38 mm 6 MHz linear probe of the ultrasound device, , the patient will be placed in the lateral decubitus position and SAP block will be applied to the serratus anterior muscle fascia using 20 ml of 0.25% bupivacaine solution.
  Interventions: Procedure: serratus anterior plane block and pectointercostal plane block in breast surgery
- serratus anterior plane block to the pecto intercostal plane block will be applied. (Other): SAP block will be applied to the patient's serratus anterior fascia using 20 ml of 0.25% bupivacaine solution. Then, PIFB will be applied to the patient's parasternal region using 10 ml of 0.25% bupivacaine solution.
  Interventions: Procedure: serratus anterior plane block and pectointercostal plane block in breast surgery

INTERVENTIONS:
Procedure: serratus anterior plane block and pectointercostal plane block in breast surgery — Serratus anterior plane block and pecto intercostal plane block will be performed as a single injection using 0.25% bupivacaine and with the same practitioner.

SUMMARY:
the study is a clinical study that will be conducted on women between the ages of 18 and 75 who are scheduled for breast surgery. We aimed to compare the postoperative pain management effect of adding the pecto intercostal fascial plane block to the serratus anterior plane block.

DETAILED DESCRIPTION:
Patients between the ages of 18-75 who are scheduled for breast surgery, who are in American Society of Anesthesiologists (ASA) class I-III groups, who are not pregnant or suspected of being pregnant, and who approve the informed consent form will be included in the study. Patients with known local anesthetic allergy or suspected coagulopathy, injection site infection, serious neurological or psychiatric disorder, severe cardiovascular disease, liver failure, renal failure (glomerular filtration rate <15 ml/min/1.73 m2) and chronic opioid use are excluded from the study will be left.

Within the scope of this study, two different research groups were identified for which clinical research was planned. The significance level of the power analysis was determined as 0.05 and the power level was determined as 0.80. However, for this study, it was decided to consider the effect size value as 0.4, based on similar studies in the literature. It was deemed sufficient to include n = 26 cases in each group, and it was deemed appropriate to include n = 30 cases in each group, considering a 20% wastage margin. The cases will be divided into 2 groups of 30 people using the sealed envelope method. Group I will include patients who underwent SAP block under general anesthesia (Control group), and Group II will include patients who underwent SAP and PIFB block under general anesthesia (Experimental group). Demographic information (weight, height, age, body mass index, comorbidity ASA score) of all cases will be recorded. After informed consent was obtained in all cases; Standard monitoring including HR, SS, SpO2 non-invasive blood pressure, and 5-lead electrocardiography will be performed. Following anesthesia induction with midazolam 0.05 mg\kg intravenous (IV), propofol 2.5 mg\kg IV, fentanyl 2 mcg\kg IV, lidocaine 1 mg\kg IV and rocuronium 1 mg\kg IV, which the investigators routinely use in our clinic for general anesthesia. It is planned to maintain anesthesia with sevoflurane in patients whose airway is provided with a laryngeal mask, with a minimum alveolar concentration (MAC) of 1. The patient is placed in the lateral decubitus position and serratus guided by the 38 mm 6 MHz linear probe of the ultrasound device, which is routinely applied to Group I (Control group) patients in our clinic. SAP block will be applied to the anterior muscle fascia using 20 ml of 0.25% bupivacaine solution. For Group II (Experimental group) patients, SAP block will be applied to the serratus anterior muscle fascia using 20 ml of 0.25% bupivacaine solution, accompanied by the 38 mm 6 MHz linear probe of the ultrasonography device that is routinely applied in our clinic. The patient will be placed in the lateral decubitus position. Then, the patient will be placed in the supine position and 4 strokes will be applied in the parasternal region. PIFB will be applied using 10 ml of 0.25% bupivacaine solution between the pectoralis major and external intercostal muscle fasciae at the level of the intercostal space. In the intraoperative period, paracetamol 1000 mg IV and tenoxicam 20 mg IV will be administered to all patients as the investigators routinely apply. The patients' hemodynamic data and the amount of opioid used during the operation will be recorded every 30 minutes during the intraoperative period.

In the postoperative period, patients' visual pain score (VAS) and VAS score during movement will be measured at the 1st, 2nd, 4th, 8th, 12th and 24th hours. In addition, the patients' first additional analgesic time, additional analgesic requirement and consumption amount will be recorded.

It is planned to give paracetamol 4x500 mg IV as a rescue analgesic in patients with a VAS score of 4 and above in the postoperative period, and tramadol 1 mg\kg IV as a second rescue analgesic in patients whose VAS score continues to be 4 and above during their follow-up.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I-III groups,
* not pregnant or suspected of being pregnant
* approve the informed consent form will be included in the study.

Exclusion Criteria:

* Patients with known local anesthetic allergy or suspected coagulopathy,
* Infection on injection area
* Serious neurological disorder
* Psychiatric disorder
* Severe cardiovascular disease
* Liver failure
* Renal failure
* Using chronic opioid

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients' VA scores should be below 4 within 24 hours post-operatively and the need for analgesia should be reduced or absent.
Enrollment: 60 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-05-07 (Estimated)

PRIMARY OUTCOMES:
Change on analgesic needs of patients in the first 24 hours postoperatively | within posoparativ 24 hours
  Patients' visula pain score should be below 4 within 24 hours post-operatively and the need for analgesia should be reduced or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Yavaşçaoglu, prof, Study Director — Uludag University Medicine Faculty; SELCAN AKESEN, assoc.prof, Study Chair — Uludag University Medicine Faculty
Locations (1):
- ULUDAGU, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No